CLINICAL TRIAL: NCT05507125
Title: Regulation of Inflammatory Genes in Hidradenitis Suppurativa
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Nabiha Yusuf, Professor, University of Alabama at Birmingham
Other Study IDs: 300006000
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Mental Health

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: Participants without inflammatory skin disease
  Interventions: Behavioral: Mental health
- Patients with HS: Patients with HS
  Interventions: Behavioral: Mental health

INTERVENTIONS:
Behavioral: Mental health — Early life exposure to abuse and development of hidradenitis suppurativa

SUMMARY:
The purpose of this protocol is to examine the cytokine profi le of pati ents with hidradeniti s suppurati va (HS) and idemechanisms responsible for post-transcripti onal regulati on of these genes. The primary objecti ve is to determinfollowing cytokines linked to hidradeniti s suppurati va are diff erenti ally expressed in hidradeniti s pati ents versus controlalso doing a sub-study to determine the eff ect of childhood trauma on HS. The parti cipati on in the sub-study is opti onal

DETAILED DESCRIPTION:
Hidradeniti s suppurati va (HS) is a chronic infl ammatory cutaneous disease which involves the pilosebaceous-apocrwhich typically presents aft er puberty with painful nodules and abscesses which can form sinus tracts and scars in theapocrine gland-bearing sites of the body. 1 Esti mates of disease prevalence range from 0.0003% to 4%, with youngparti cularly women as the most eff ected group. Racial predilecti on has also been demonstrated, with a higher likeldisease in African American and biracial individuals when compared to whites.1 HS is an under-recognized enti ty, ontaking 7.2 years from symptom onset to formal diagnosis.2 A notable aspect of HS is the profound impact it can have oof life in pati ent's suff ering with the disease, with an increase in depression, pain, and social and work impairment.pathogenesis conti nues to be elucidated but is primarily thought to be due to follicular hyperkeratosis, leading formati on, dilati on, and rupture. This in turn causes infl ammati on, abscess and sinus tract formati on. 1, 4 Whiunderstanding of a role of tumor necrosis factor (TNF) alpha, interleukin (IL)-1, IL-17A, IL-23, C-reacti ve protein (Cinterferon (IFN) gamma have been previously shown, much is sti ll unknown of the molecular involvement of infl ammarkers in HS.1, 2, 4. Currently, management varies from topical treatment, to surgical excision, to prescribing manbiologic medicati ons used for hidradeniti s suppurati va and infl ammatory bowel disease. However, there can be vasvariability in response to these medicati ons, and a proper understanding of the infl ammatory markers involved inpathogenesis will allow for more specifi c treatment, while hopefully avoiding the adverse eff ects related to these isuppressive medicati ons. Thus, in this study we will assess the cytokines, TNF-alpha, IFN-gamma, IFN-alpha, IFN-beta, IIL-12, IL-23, IL-17A, and study their regulati on in HS lesions of pati ents, with the ulti mate goal of identi fying potenti al tafuture therapies and interventi ons.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hidradenitis suppurativa
* Not Pregnant

Exclusion Criteria:

* Mild/general dermatological issues like moles, other cosmetic issues
* Patients with hidradenitis suppurativa, psoriasis, roasacea, atopic dermatitis and other inflammatory skin disease
* Pregnant

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hidradenitis suppurativa is an autoinflammatory skin disorder.They are difficult-to-heal and often scar. Hidradenitis suppurativa also has a significant psychological impact, and many patients suffer depression, anxiety, and impaired body-image. A hallmark of hidradenitis suppurativa is increased levels of biomarkers, which are molecules found in blood, other body fluids, or tissues that can be a sign of a normal or abnormal process. In hidradenitis suppurativa, these biomarkers are called "cytokines" and their job is to trigger the disease and make it worse.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Inflammatory biomarkers | 24 hours after application
  Inflammatory biomarkers

SECONDARY OUTCOMES:
Cytokines | 24 hours after application
  Cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Nabiha Yusuf, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Whitaker Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided